CLINICAL TRIAL: NCT06598800
Title: A Phase 1 Study Investigating the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of BG-T187, an EGFR×MET Trispecific Antibody, Alone and in Combination With Other Therapeutic Agents in Patients With Advanced Solid Tumors
Brief Title: Study of BG-T187 Alone and in Combination With Other Therapeutic Agents in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BG-T187-101; 2024-514944-10-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumors; First-in-human; BG-T187; EGFR; c-MET

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1a: Part A: Monotherapy Dose Escalation with Intravenous Administration (Experimental): Sequential cohorts of increasing dose levels of BG-T187 will be evaluated as monotherapy.
  Interventions: Drug: Drug: BG-T187
- Phase 1a: Part B: Monotherapy Dose Escalation with Subcutaneous Administration (Experimental): Sequential cohorts of increasing dose levels of BG-T187 will be evaluated as monotherapy.
  Interventions: Drug: Drug: BG-T187
- Phase 1a Part C: Safety Expansion (Experimental): BG-T187 dose levels that have been determined to be safe and tolerable in Part A will be investigated.
  Interventions: Drug: Drug: BG-T187
- Phase 1b: Monotherapy Dose Expansion with Subcutaneous Administration (Experimental): Participants will receive BG-T187 monotherapy at the recommended dose(s) for expansion (RDFE) determined in Phase 1a.
  Interventions: Drug: Drug: BG-T187
- Phase 1b: Combination Therapy: BG-T187 + Other Therapeutic Agents (Experimental): Participants will receive BG-T187 in combination with Other Therapeutic Agents.
  Interventions: Drug: Drug: BG-T187; Drug: Other Therapeutic Agents

INTERVENTIONS:
Drug: Drug: BG-T187 — administered subcutaneously
Drug: Other Therapeutic Agents — administered intravenously
  Arms: Phase 1b: Combination Therapy: BG-T187 + Other Therapeutic Agents

SUMMARY:
This is a first-in-human (FIH), Phase 1a/1b, open-label, multicenter, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary antitumor activity of BG-T187 alone and in combination with other therapeutic agents in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide a signed and dated written informed consent prior to any study-specific procedures, sampling, or data collection.
2. Participants must be ≥ 18 years of age or the legal age of consent in the jurisdiction in which the study is taking place.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
4. Participants with selected histologically or cytologically confirmed advanced, metastatic, and unresectable solid tumors who have been previously treated.
5. ≥ 1 measurable or nonmeasurable lesion as assessed by RECIST v1.1. for Phase 1a Part A; ≥ 1 measurable lesion per RECIST v1.1. for Phase 1a Part B and Phase 1b.
6. Adequate organ function.

Exclusion Criteria:

1. Prior severe allergic reactions or hypersensitivity to the active ingredient and excipients of BG-T187 or other monoclonal antibodies.
2. Spinal cord compression, active leptomeningeal disease, or uncontrolled, untreated brain metastasis.
3. Any malignancy ≤ 3 years before the first dose of study drug(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast).
4. History of interstitial lung disease (ILD) or noninfectious pneumonitis requiring steroids or other immune suppressive agents ≤ 2 years before the first dose of the study drug, or with current ILD/noninfectious pneumonitis, or where suspected ILD/noninfectious pneumonitis cannot be ruled out by imaging during screening.
5. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage (recurrence ≤14 days after intervention).
6. Active hepatitis C.
7. Infection (including tuberculosis infection, or other) requiring systemic (oral or intravenous) antibacterial, antifungal, or antiviral therapy ≤ 14 days before the first dose of study drug(s).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Approximately 2 years
  Number of participants with AEs including serious adverse events (SAEs), defined as any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease temporally associated with the use of study drugs, whether considered related to study drugs or not as graded by the National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI CTCAE) V5.0/American Society for Transplantation and Cellular Therapy (ASTCT) for cytokine release syndrome [CRS] and immune effector cell associated neurotoxicity syndrome [ICANS]); and adverse events meeting protocol-defined dose-limiting toxicity (DLT) criteria
Phase 1a: Maximum Administered Dose (MAD) or Maximum Tolerated Dose (MTD) of BG-T187 | Approximately 2 years
  MTD or MAD is defined as the highest dose evaluated for which the estimated toxicity rate is closest to the target toxicity rate of 30% or the highest dose administered, respectively.
Phase 1a: Recommended Dose(s) for Expansion (RDFE[s]) of BG-T187 | Approximately 2 years
  RDFE(s) is determined based on the MAD or MTD, taking into consideration the long-term tolerability, pharmacokinetics (PK), preliminary antitumor activity, and any other relevant data, as available
Phase 1b: Overall Response Rate (ORR) | Approximately 2 years
  ORR is defined as the percentage of participants with confirmed best overall response (BOR) complete response (CR) or partial response (PR) as determined by investigators per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Phase 1b: Recommended Phase 2 dose (RP2D) of BG-T187 alone and in combination with other therapeutic agents | Approximately 2 years
  R2PD is determined based on safety, tolerability, PK, preliminary antitumor activity, and other relevant data, as available

SECONDARY OUTCOMES:
Phase 1a: ORR | Approximately 2 years
  ORR is defined as the percentage of participants with confirmed BOR, CR or PR as determined by investigators per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Phase 1a and 1b: Duration of Response (DOR) | Approximately 2 years
  DOR is defined as the time from the first objective response until the first documentation of disease progression after treatment initiation or death, whichever comes first, as determined by investigators per RECIST v1.1
Phase 1a and 1b: Disease Control Rate (DCR) | Approximately 2 years
  DCR is defined as the percentage of participants with the BOR of confirmed CR, PR, or stable disease, as determined by investigators per RECIST v1.1
Phase 1b: Progression Free Survival (PFS) | Approximately 2 years
  PFS is defined as the time from the date of the first administration of study drug to the date of the first documentation of disease progression or death due to any cause, whichever occurs first, as determined by investigators per RECIST v1.1
Phase 1a: Maximum observed plasma concentration (Cmax) of BG-T187 | From Cycle 1 to Cycle 3 (each cycle is 28 days)
Phase 1a: Area Under the Plasma Concentration-time Curve (AUC) of BG-T187 | From Cycle 1 to Cycle 3 (each cycle is 28 days)
Phase 1a: Terminal Half-Life (t1/2) of BG-T187 | From Cycle 1 to Cycle 3 (each cycle is 28 days)
Phase 1a: Time to maximum plasma concentration (Tmax) of BG-T187 | From Cycle 1 to Cycle 3 (each cycle is 28 days)
Phase 1a and 1b: Number of participants with anti-drug antibodies (ADAs) to BG-T187 | From Cycle 1 Day 1 up to 30 days after last dose (approximately 2 years)
Phase 1b: Number of Participants with AEs and SAEs | Approximately 2 years
  Number of participants with AEs including serious adverse events (SAEs), defined as any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease temporally associated with the use of study drugs, whether considered related to study drugs or not as graded by the National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI CTCAE) V5.0/American Society for Transplantation and Cellular Therapy (ASTCT)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (25):
- United States (4):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
  - Next Virginia, Fairfax, Virginia
  - Washington University, St Louis, Division of Oncology, Madison, Wisconsin
- Australia (4):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Macquarie University, North Ryde, New South Wales
  - Cabrini Hospital Malvern, Malvern East, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- China (10):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The Sixth Affiliated Hospital, Sun Yat Sen University, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Linyi Peoples Hospital, Linyi, Shandong
  - The First Affiliated Hospital, Zhejiang University School of Medicinezhijiang Branch, Hangzhou, Zhejiang
- South Korea (7):
  - Seoul National University Bundang Hospital, BundangGu SeongnamSi, Gyeonggi-do
  - The Catholic University of Korea, St Vincents Hospital, PaldalGu SuwonSi, Gyeonggi-do
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St Marys Hospital, SeochoGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/